CLINICAL TRIAL: NCT01747824
Title: Stress Biomarkers Among Patients Undergoing Treatment for Excited Delirium and Severe Pain in the Emergency Department
Acronym: Agitation
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 12-3478
Record Dates: First submitted 2012-12-04; First posted 2012-12-12 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Agitation; Excited Delirium; Pain
Keywords: agitation; excited delirium; pain; unexplained-in-custody-death; UICD; visual analog scale; VAS; altered mental status; AMS
MeSH Terms: conditions — Psychomotor Agitation; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Agitation Group: Patients that are evaluated to have an altered mental status score greater than 1 will be enrolled in the Agitation Group.
- Pain Group: Patients that report severe pain secondary to a long bone fracture or dislocation and report a visual analog scale pain score greater than 7 will be enrolled in the Pain Group.

SUMMARY:
The purpose of this project is to determine the levels of stress biomarkers associated with severe pain, agitation from intoxication or psychosis, and excited delirium at various levels of the disease in order to compare them to pre-clinical models of law enforcement encounters. We hypothesize that the serum catecholamines and markers of metabolic acidosis will worsen with the duration and severity of agitation among agitated patients and will not worsen among patients with severe pain who are not agitated.

Specific Aims

* To assess the prevalence of patients undergoing treatment for agitation from any cause requiring restraint or sedation.
* To assess the prevalence of excited delirium in the emergency department.
* To determine the difference in serum total catecholamines, serum dopamine, serum epinephrine, serum norepinephrine, heart rate, systolic blood pressure, mean arterial pressure, mortality, and disposition among patients with agitation requiring restraint, including excited delirium and patients with severe pain from extremity fractures.
* To describe changes in stress biomarkers among patients with changing levels of agitation as determined by the Altered Mental Status scale.

DETAILED DESCRIPTION:
In this study, we propose to study Emergency Department patients under physiologic stress from severe pain, agitation, drug overdose, and excited delirium in order to compare markers of acidosis in patients at risk for unexplained-in-custody-death (UICD) in order to determine the relationship of these markers to what has been found in simulated law enforcement encounters. This information will help clarify the levels of stress associated with arrest and restraint conditions, allowing us to determine what aspects and levels of stress may be associated with the fatal mechanisms of UICD, and to identify markers that would inform death investigators of the mechanism of UICD. At the conclusion of this project, we will be able to report details explaining the relationship of the physiologic and metabolic effects of stress from restraint in excited delirium to other peri-arrest conditions and our previous work in simulated law enforcement encounters.

ELIGIBILITY:
Agitation Group Inclusion Criteria:

* Patients with agitation as defined by an Altered Mental Status Score of >1, and who are in restraints or are given sedatives for treatment of agitation.

Agitation Group Exclusion Criteria:

* Less than 18 years of age
* Suspected or confirmed pregnancy

Pain Group Inclusion Criteria:

* Patients with an extremity fracture who report their pain as severe.

Pain Group Exclusion Criteria:

* Less than 18 years of age
* Suspected or confirmed pregnancy
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing treatment for acute agitation in the emergency department of an urban Level 1 Trauma Center.
Sampling Method: Probability Sample
Enrollment: 1322 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Altered Mental Status Score | Assessed every five minutes, from enrollment until discharge from the emergency department, an expected average time of 4 hours
Change in Visual Analog Scale Pain Score | Assessed every five minutes, from enrollment until discharge from the emergency department, an expected average time of 4 hours
Change in Serum Total Catecholamines | Assessed every 30 minutes, from enrollment until discharge from the emergency department, an expected average time of 4 hours
  Serum dopamine, serum epinephrine, and serum norepinephrine.

SECONDARY OUTCOMES:
Length of Hospital Stay | Assessed at time of discharge from the hospital, an expected average of 4 hours post enrollment.
Mortality | Observed for 1 year post study enrollment
Complications | Observed for 1 year post study enrollment
Change in Heart Rate | Observed from time of enrollment until discharge from the emergency department, an expected average time of 4 hours
Change in Systolic Blood Pressure | Observed from time of enrollment until discharge from the emergency department, an expected average time of 4 hours
Change in Mean Arterial Pressure | Observed from time of enrollment until discharge from the emergency department, an expected average time of 4 hours
Disposition | Assessed at discharge from the emergency department, an expected average of 4 hours post enrollment.
Change in Body Temperature | Observed from time of enrollment until discharge from the emergency department, an expected average time of 4 hours
Change in end tidal carbon dioxide | Assessed from time of enrollment until discharge from the emergency department, an expected average time of 4 hours
Change in Oxygen Saturation | Observed from time of enrollment until discharge from the emergency department, an expected average time of 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: James R Miner, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Miner JR, Klein LR, Cole JB, Driver BE, Moore JC, Ho JD. The Characteristics and Prevalence of Agitation in an Urban County Emergency Department. Ann Emerg Med. 2018 Oct;72(4):361-370. doi: 10.1016/j.annemergmed.2018.06.001. Epub 2018 Jul 19. PMID 30031556